CLINICAL TRIAL: NCT06002724
Title: Feasibility Study of Peripheral Venous Cannulation Pain in Predicting Acute Pain After
Brief Title: Feasibility Study of Peripheral Venous Cannulation Pain in Predicting Acute Pain After Total Knee Arthroplasty
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: taoliqin0730
Record Dates: First submitted 2023-08-16; First posted 2023-08-21 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Venous Cannulation Pain; Total Knee Arthroplasty; Movement-evoked Pain; Acute Pain
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 0

INTERVENTIONS:
Other:

SUMMARY:
The goal of this prospective observational study is to explore the feasibility of preoperative peripheral venous cannulation pain score in predicting acute pain after total knee arthroplasty, including resting pain and movement-evoked pain.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing the first unilateral total knee arthroplasty surgery under general anesthesia combined with nerve block ;
2. Age : 18 years old ≤ age ≤ 80 years old ;
3. ASA grade I-II ;
4. Informed consent was signed by patients or immediate family members before operation.

Exclusion Criteria:

1. There are known pain abnormalities, mental disorders, cognitive dysfunction ;
2. patients with long-term use of opioids and a history of drug dependence ;
3. patients with alcohol dependence ;
4. the patient refused to use the analgesic pump ;
5. Difficult to understand the VAS score ;
6. body mass index ≥ 40 ;
7. hand nerve abnormalities, hand loss ;
8. plan postoperative ICU patients ;
9. In other cases, the researchers believe that is not suitable for this researcher.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing unilateral total knee arthroplasty for the first time under general anesthesia combined with nerve block
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2023-08-30 (Estimated); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
postoperative resting pain and movement-evoked pain | one hour、the first day and the second day after operation
  visual analogue scale（VAS) of one hour、the first day and the second day after operation

IPD SHARING:
Plan to Share IPD: No